CLINICAL TRIAL: NCT00676234
Title: Recombinant Human Erythropoietin Use in ICU Patients: Does it Prevent Acute Renal Failure?
Brief Title: Recombinant Human Erythropoietin Use in Intensive Care Unit (ICU) Patients: Does it Prevent Acute Renal Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Dr P. Saudan, Nephrology Unit
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-11021991
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Acute Renal Failure
Keywords: erythropoietin
MeSH Terms: conditions — Acute Kidney Injury | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Administration of intravenous rhu Epo on Day 0
  Interventions: Drug: epoetinum

INTERVENTIONS:
Drug: epoetinum — Administration of intravenous rhu Epo on Day 0 20000 IU rhu Epo (20 patients) administered by the i.v. route 40000 IU rhu Epo (20 patients) administered by the i.v. route
  Other Names: Eprex
  Arms: 2

SUMMARY:
Pilot study aiming to assess the effect of two doses of rhu EPO on urine NGAL concentration and on serum cystatin C and creatinine levels in critically ill patients at risk of ARF.

DETAILED DESCRIPTION:
Research plan Open-label randomized trial Twelve months duration trial Setting: Medical and Surgical Intensive Care Unit of the University Hospitals of Geneva Start of trial: Mid-May 2008

Patients randomly allocated to 2 treatment groups (20 patients per group), or a control group (40 patients):

* Group 1: control group (40 patients)
* Group 2 : 20000 IU rhu Epo (20 patients) administered by the i.v. route
* Group 3 : 40000 IU rhu Epo (20 patients) administered by the i.v. route

3.2. Trial design Day 0 Consent form signed Patients randomly allocated to control or treatment groups (20000 and 40000 IU) Serum Cystatin C determination Serum Creatinine determination Urinary NGAL determination Administration of intravenous rhu Epo on Day 0 or no Epo (control group) Day 2 At 48 hr after rhu EPO injection, samples will be taken for

* Serum Cystatin C determination
* Serum Creatinine determination
* Urinary NGAL determination Day 4 At 96 hr after rhu EPO injection, samples will be taken for
* Serum Cystatin C determination
* Serum Creatinine determination
* Urinary NGAL determination

Stopping rules

The trial for an individual subject, parts of the trial or the entire trial will be stopped when:

* at Day 4 for an individual subject
* after enrollment of 80 patients

Treatment The treatment will consist of intravenous (i.v.) injections of recombinant human erythropoietin (r-hu-EPO). The trial medication will be provided by JANSSEN-CILAG AG. The brand name is EPREX® which is epoietinum-alpha in sterile buffered solution for i.v. or s.c. injection.

Patient group 1 will not receive EPO treatment. Patient group 2 will receive 20'000 U of rhu EPO and patient group 3 will receive 40'000 U of rhu EPO (i.v. route).

ELIGIBILITY:
Inclusion Criteria:

* Patients at risks for acute tubular necrosis (patients with mechanical ventilation, patients with sepsis, in the post-operative state, with hemodynamic impairment or with previous chronic renal failure.
* Consent form signed

Exclusion Criteria:

* Patients with malignant hypertension
* Patients with systolic BP > 150 mmHg at enrollment
* Patients with Hb level > 120g/L
* Patients with acute coronaropathy
* Pregnancy
* Patients with urine output < 600 ml/12 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
mean change (%) from baseline in urinary NGAL concentration at 96 hr after rhu EPO injection | 4 days

SECONDARY OUTCOMES:
mean change (%) from baseline in serum Cystatin C concentration at 96 hr after rhu EPO injection | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Saudan, Dr, Principal Investigator — Nephrology Unit Geneva University Hospitals
Locations (1):
- Nephrology Unit, Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879
- [Derived] de Seigneux S, Ponte B, Weiss L, Pugin J, Romand JA, Martin PY, Saudan P. Epoetin administrated after cardiac surgery: effects on renal function and inflammation in a randomized controlled study. BMC Nephrol. 2012 Oct 3;13:132. doi: 10.1186/1471-2369-13-132. PMID 23033926